CLINICAL TRIAL: NCT04160000
Title: A Phase 4, Randomized, Open Label, Multicenter Prospective Comparative Study To Evaluate The Treatment Of Atrial Fibrillation In Preserved Cardiac Function Heart Failure
Brief Title: Treatment Of Atrial Fibrillation In Preserved Cardiac Function Heart Failure
Acronym: TAP-CHF
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Electrophysiology Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EPRF - 2019 - 11
Record Dates: First submitted 2019-11-06; First posted 2019-11-12 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-05

CONDITIONS: Atrial Fibrillation; Heart Failure; Diastolic Heart Failure
Keywords: Atrial fibrillation; Heart failure; Diastolic heart failure; Catheter Ablation; Antiarrhythmic Drugs
MeSH Terms: conditions — Atrial Fibrillation; Heart Failure; Heart Failure, Diastolic | interventions — Catheter Ablation; Anti-Arrhythmia Agents

STUDY DESIGN:
Intervention Model Description: This is a prospective pilot study utilizing a randomized comparative sequential evaluation of two therapeutic approaches in two consecutive phases. Phase 1 will examine an initial catheter ablation strategy versus an initial antiarrhythmic drug (AAD) therapy strategy for safety and efficacy in patients with atrial fibrillation with preserved systolic cardiac function, heart failure hospitalization in the past year or one or more documented HF events.
  Phase 2 will examine optimized rhythm control therapy with and without wireless pulmonary artery pressure hemodynamic monitoring for HF therapy optimization in the same patients as in Phase 1 with documented atrial fibrillation with preserved systolic cardiac function, prior HF hospitalization and class III heart failure.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- Phase 1 Catheter Ablation (Active Comparator): Patients with atrial fibrillation and heart failure with preserved systolic function will be enrolled after informed consent. They randomly assigned to catheter ablation as one arm. They will undergo a catheter ablation procedure within 14 days of randomization. This procedure will include isolation of all four pulmonary veins in the antrum using catheter delivered radiofrequency current, cryothermal or laser ablation energy with standard FDA approved ablation catheter systems used in atrial fibrillation ablation. Patients will be monitored for a minimum period of 9 months after the catheter ablation intervention.
  Interventions: Device: Catheter ablation
- Phase 1 Antiarrhythmic drug therapy (Active Comparator): Patients with atrial fibrillation and heart failure with preserved systolic function will be enrolled after informed consent. They will be randomly assigned to antiarrhythmic drug therapy for Rate or Rhythm control in this arm. They will undergo drug dose titration within 14 days of randomization. . Patients will be monitored for a minimum period of 9 months after the AAD therapy initiation
  Interventions: Drug: Rate or Rhythm control antiarrhythmic drugs for atrial fibrillation
- Phase 2 Guided Heart Failure Therapy (Active Comparator): Patients with atrial fibrillation and heart failure with preserved systolic function will be enrolled after informed consent and completion of Phase 1. They will be randomly assigned to insertion of an implantable hemodynamic monitor in this arm and heart failure therapy guided by wireless hemodynamic monitoring. Patients will be monitored for a minimum period of 9 months after the implantable hemodynamic monitor insertion on guided drug therapy
  Interventions: Device: Insertion of CardioMems Hemodynamic monitor
- Phase 2 Empiric Heart Failure Therapy (Active Comparator): Patients with atrial fibrillation and heart failure with preserved systolic function will be enrolled after informed consent and completion of Phase 1. They will be randomly assigned to heart failure management with empirical selection of heart failure therapy. Patients will be monitored for a minimum period of 9 months after the initiation of empirically selected heart failure drug therapy
  Interventions: Drug: Empiric heart failure drug therapy

INTERVENTIONS:
Device: Catheter ablation — Delivery of physical energy from external energy source via percutaneously inserted electrophysiologic catheter to destroy heart tissue in the human atrium and adjoining vasculature
  Other Names: Ablation
  Arms: Phase 1 Catheter Ablation
Drug: Rate or Rhythm control antiarrhythmic drugs for atrial fibrillation — Administration of antiarrhythmic drug to achieve either rate control or restoration of sinus rhythm for management of atrial fibrillation
  Other Names: Antiarrhythmic Drug
  Arms: Phase 1 Antiarrhythmic drug therapy
Device: Insertion of CardioMems Hemodynamic monitor — Insertion of wireless hemodynamic monitor to provide hemodynamic data to guide heart failure therapy to achieve heart failure improvement.
  Other Names: IPM
  Arms: Phase 2 Guided Heart Failure Therapy
Drug: Empiric heart failure drug therapy — Administration of heart failure drug therapy based on clinical evaluation to achieve heart failure improvement.
  Other Names: HFDrug
  Arms: Phase 2 Empiric Heart Failure Therapy

SUMMARY:
Heart failure (HF) with preserved left ventricular function (pEF) is difficult clinical syndrome to treat effectively with few evidence based therapies. Atrial fibrillation (AF) is now an important co-morbidity being observed in 43% of patients with HFpEF. Rhythm control has not been studied in this population. Catheter ablation and antiarrhythmic drugs are rhythm control therapies that have been used for treatment of AF without HF or HF with reduced systolic function but have not been widely applied in HFpEF. No controlled comparative evaluation has been performed in HFpEF.

The introduction of wireless pulmonary artery hemodynamic monitoring has permitted optimization of HF therapy in patients with chronic HF with reduced and preserved EF. Reduction in HF hospitalizations has been observed in post hoc analyses of HFpEF patients but has not been systematically applied in AF patients with HFpEF.

In this study, we propose to study both rhythm control and optimized HF therapeutic approaches in an AF with HFpEF study population in a pilot study using a sequential two phase randomized controlled clinical trial design.

DETAILED DESCRIPTION:
This is a prospective pilot study utilizing a randomized comparative sequential evaluation of these two therapeutic approaches in two consecutive phases:

Phase 1 will examine an initial catheter ablation strategy versus an initial antiarrhythmic drug (AAD) therapy strategy for safety and efficacy in patients with atrial fibrillation with preserved systolic cardiac function, heart failure hospitalization in the past year or one or more documented HF events.

Phase 2 will examine optimized rhythm control therapy with and without wireless pulmonary artery pressure hemodynamic monitoring for HF therapy optimization in the same patients as in Phase 1 with documented atrial fibrillation with preserved systolic cardiac function, prior HF hospitalization and class III heart failure.

This is an open label two phase study in which patients will be randomized in a 1:1 ratio to either ablation or AAD with a pilot phase 1 that will consist to 100 patients enrolled at 10 centers. They will be followed for a minimum of 6 months, after a three month blanking period, for event rates of the primary endpoint as well as safety and efficacy. Phase 2 will randomize patients completing Phase 1 to hemodynamic monitoring with a wireless pulmonary artery sensor insertion and guided HF therapy or empiric standard of care HF therapy. They will be followed for a minimum of 6 months, after a three month blanking period for optimization of rhythm and HF therapies.

This study is a sequential randomized, open label, active-controlled trial, designed to compare a composite clinical outcomes endpoint of heart failure hospitalization and/or cardiovascular mortality among these patients randomized to each of these treatment strategies. This endpoint will be employed in both pilot trial phases to assess event rates, as well as safety endpoints. This data will form the basis of a larger pivotal trial

ELIGIBILITY:
Inclusion Criteria: Patient with symptomatic Heart Failure with preserved systolic cardiac function & paroxysmal or persistent atrial fibrillation who meet the following criteria

1. Subjects must be willing and able to give written informed consent
2. Outpatients ≥ 50 years of age, male or post- menopausal female patients; premenopausal female patients who are on and will maintain continuous birth control therapy during the study.
3. Subjects must have documented HFpEF & paroxysmal or persistent AF and satisfy one of the following inclusion criteria a) Consecutive patients with AF, symptomatic heart failure requiring diuretic therapy for at least 30 days prior to study entry b) Hospitalization for HF and/or AF in the past 12 months prior to catheter ablation with documented NT-pro BNP >200pg/ml for patients not in AF or > 600 pg/ml for patients in AF on screening ECG or NYHA class 2, 3 or ambulatory class 4 heart failure documented NT-pro BNP >300pg/ml for patients not in AF or > 900 pg/ml for patients in AF on screening ECG c).Evidence of structural heart disease defined as by at least 1 of the following echocardiography findings (any local measurement made during the screening epoch or within the 6 months prior to screening visit): 1) LA enlargement defined by at least 1 of the following: LA width (diameter) >3.8 cm or LA length >5.0 cm or LA area >20 cm2 or LA volume >55 ml or LA volume index >29 ml/m2 2) LVH defined by septal thickness or posterior wall thickness >1.1 cm d).Left ventricular ejection fraction > 45% using standard imaging techniques at enrollment for study or in prior 6 months e).ECG documented paroxysmal or persistent atrial fibrillation f).Patients are candidates for a clinically indicated catheter ablation procedure, and Rate or Rhythm control antiarrhythmic drug therapy
4. Patients should be on one or more standard heart failure drug therapy (ies) for heart failure with preserved cardiac function for at least 30 days
5. Written informed consent for the clinically indicated study procedures
6. Patients must be candidates for long-term OAC therapy based on clinical practice guidelines for treatment of AF. Guidelines for GFR as established for DOACSs will be applicable to all subjects.

Exclusion Criteria:

1. Patients with HFpEF who were not on any drug therapy for HF or have uncontrolled hypertension defined as systolic BP >180 mm Hg at screening or >150 mm Hg on three or more antihypertensive drugs
2. Patients with QRS duration of >120 ms and intraventricular conduction defects who are or maybe candidates for or have received ventricular resynchronization therapy
3. Recent (<1 month) myocardial infarction or acute coronary syndrome
4. Recent (<3 months) coronary revascularization procedures
5. Documented LA thrombus on TEE or any LVEF measurement <40%
6. Patients who are not candidates for Rate or Rhythm control drug therapy for AF
7. Dilated cardiomyopathy due to potentially reversible cause e.g. myocarditis
8. Contraindications to anticoagulant therapy or adverse event with prior Warfarin or DOAC therapy
9. Creatinine clearance <30ml/min or >95ml/min
10. Advanced hepatic disease, pulmonary disease clinically significant congenital heart disease, clinically significant pericardial constriction, hypertrophic cardiomyopathy, infiltrative cardiomyopathy, decompensated valvular heart disease likely to require surgical or percutaneous intervention during the trial
11. Recent stroke (<3 months) or thromboembolic event, transient ischemic attack or carotid angioplasty in the prior 3 months
12. Recent (<3 months) intracranial or other major bleeding event
13. Candidates for heart or any other organ transplantation or left ventricular assist devices, recent (< 3 months) valve or other cardiac surgery
14. Patients requiring ACE inhibitor or ARB drug therapy for any reason
15. History of hypersensitivity to antiarrhythmic drugs
16. Patients with other clinically significant medical condition that precludes study participation
17. Patients with life expectancy < 1 year
18. Premenopausal female patients, who are not on continuous birth control therapy or are likely to discontinue it at any time during the entire duration of study enrollment.
19. Pregnant or nursing lactating mothers or women of childbearing potential who are not on effective contraceptive therapy
20. Patients who have been noncompliant with medical regimens or have social or other issues precluding regular follow up, history of alcohol or drug abuse in past 12 months.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2020-07-26 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Time to Composite of Heart failure hospitalizations and/or Cardiovascular mortality | From date of randomization until the date of first documented heart failure hospitalization or date of death from cardiovascular causes, whichever came first, assessed up to 12 months
  Time to either first of Heart failure hospitalization and/or mortality due to cardiovascular etiology

SECONDARY OUTCOMES:
All cause Mortality | From date of randomization until the date of death from any cause, assessed up to 12 months
  Time to mortality due to any cause
MACE events | From date of randomization until the date of first documented major adverse cardiovascular event, assessed up to 12 months
  Time to major adverse cardiovascular event
Cardiovascular Hospitalization | From date of randomization until the date of first documented hospitalization due to cardiovascular causes , assessed up to 12 months
  Time to first hospitalization due to cardiovascular causes

CONTACTS AND LOCATIONS:
Overall Officials: Sanjeev Saksena, MD, Study Chair — Electrophysiology Research Foundation; Andrea Natale, MD, Study Director — Electrophysiology Research Foundation
Locations (9):
- United States (7):
  - Northern Arizona Health Care, Flagstaff, Arizona
  - St. Bernards Heart and Vascular Center, Jonesboro, Arkansas
  - South Denver Cardiology, Littleton, Colorado
  - Kansas City Heart Rhythm Institute, Overland, Missouri
  - Electrophysiology Research Foundation, Warren Township, New Jersey
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - TCAI at St. David's Hospital, Austin, Texas
- Peter Osypka Herzzentrum, Munich, Bavaria, Germany
- Hopitaux Universitaires de Geneve, Geneva, Canton of Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Saksena S, Slee A. Atrial fibrillation and its pernicious role in heart failure with preserved ejection fraction: a new frontier in interventional electrophysiology. J Interv Card Electrophysiol. 2018 Mar;51(2):89-90. doi: 10.1007/s10840-018-0341-3. No abstract available. PMID 29480345
- [Background] Cikes M, Claggett B, Shah AM, Desai AS, Lewis EF, Shah SJ, Anand IS, O'Meara E, Rouleau JL, Sweitzer NK, Fang JC, Saksena S, Pitt B, Pfeffer MA, Solomon SD. Atrial Fibrillation in Heart Failure With Preserved Ejection Fraction: The TOPCAT Trial. JACC Heart Fail. 2018 Aug;6(8):689-697. doi: 10.1016/j.jchf.2018.05.005. Epub 2018 Jul 11. PMID 30007557
- [Background] Slee A, Saad M, Saksena S. Heart failure progression and mortality in atrial fibrillation patients with preserved or reduced left ventricular ejection fraction. J Interv Card Electrophysiol. 2019 Sep;55(3):325-331. doi: 10.1007/s10840-019-00534-x. Epub 2019 Mar 18. PMID 30887281
- [Background] Slee A, Saksena S. Impact of initial heart failure emergence on clinical outcomes of atrial fibrillation patients in the AFFIRM trial. Am Heart J. 2020 Feb;220:1-11. doi: 10.1016/j.ahj.2019.10.005. Epub 2019 Oct 28. PMID 31756389